CLINICAL TRIAL: NCT02408328
Title: Management of Apnea in Late Preterm and Term Infants
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Transition to new position
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Rhein, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00015842
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea | interventions — caffeine citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient Observation (Active Comparator): Continued inpatient monitoring of apnea, bradycardia, and/or desaturation until an event free period of time (5 days per the current standard of care at each participating institution) has been established and deemed appropriate for discharge home per the discretion of the responsible provider.
  Interventions: Other: Continued inpatient monitoring until apnea resolution
- Caffeine and Outpatient Monitoring (Active Comparator): Patients will receive a loading dose of caffeine on day 1 with a daily maintenance dose thereafter. Infants will then receive continued inpatient monitoring of apnea/bradycardia/desaturation until an event free period of time has been established and deemed appropriate for discharge home per the discretion of the responsible provider. Infants discharged home on caffeine therapy will receive instructions regarding use of a home monitor. Follow up in the pulmonary clinic will be arranged at 42-43 weeks gestational age. At 43 weeks corrected gestational age, caregivers will be instructed to discontinue caffeine therapy. An outpatient recorded oximetry study will be arranged at least 1 week after discontinuation of caffeine therapy. Home pulse oximetry monitoring will be discontinued if no significant events, as previously defined, are recorded.
  Interventions: Drug: Caffeine citrate; Device: Home monitor

INTERVENTIONS:
Drug: Caffeine citrate — Loading dose and continues use of caffeine until 44 weeks postmenstrual age
  Arms: Caffeine and Outpatient Monitoring
Device: Home monitor — Use of home monitor until 44 weeks postmenstrual age
  Arms: Caffeine and Outpatient Monitoring
Other: Continued inpatient monitoring until apnea resolution — Continued inpatient monitoring until apnea resolution
  Arms: Inpatient Observation

SUMMARY:
Apnea is a common discharge-delaying diagnosis in the Newborn Intensive Care Unit. While it is relatively more common in extremely premature infants, it also occurs frequently in late preterm and even full term infants. Since the majority of all births include late preterm infants and full term infants, the absolute number of late preterm and full term infants with apnea remains significant. Evidence-based guidelines for the management of apnea in such infants do not exist. Current management falls into two distinct but very different categories. This study will compare these two distinct management strategies.

Our study will be a prospective, randomized pilot trial to provide data regarding (a) feasibility for recruitment and study protocols and (b) provide preliminary data regarding efficacy of both treatment arms.

Our primary objective will be to test the hypothesis that early discharge and outpatient monitoring of late preterm and term infants with apnea of prematurity results in decreased length of hospital stay, is safe, and results in improved patient satisfaction, as assessed by the PedsQL questionnaire and Impact on Family Scale.

Our study population will include infants who meet the following criteria: (1) Born at greater than or equal to 34 0/7 weeks gestation; (2) Are assigned a diagnosis of apnea, bradycardia, and/or oxygen desaturations by the primary clinical team; (3) Have met all other discharge criteria (i.e. feeding maturity, temperature regulation, etc.) so that apnea/bradycardia/desaturation remains the final discharge issue for at least 7 days.

Infants enrolled in this research study will be randomized to in hospital observation versus early discharge home with caffeine and a home monitor. Neither strategy is experimental as both are currently utilized by neonatologists locally and nationally. A direct comparison of the two treatments, however, has never been undertaken in a study. If an infant is assigned to the in hospital group, they will remain in the hospital until an apnea free period of at least 5 consecutive days has been established. Outpatient follow up will occur per unit standard and typically includes a nursing visit and a doctor visit within 2-3 days of discharge. Caregivers will be asked to complete 3 brief questionnaires at enrollment, at 1 month after hospital discharge, and at 6 months of age. Each questionnaire will ask about topics such as satisfaction with hospital stay, quality of life, and numbers of acute care visits and/or rehospitalizations. Alternatively, if an infant is assigned to the early discharge group, caffeine will be given to the infant and if after a 3 day period no further apnea is noted the infant will be discharged home with continued daily caffeine therapy by mouth as well as a home monitor. Caffeine is a very commonly used drug in neonates and has an excellent safety profile. Side effects are minimal and may infrequently consist of gastroesophageal reflux. All caregivers will receive training on the use of a home monitor. Initial outpatient follow up will occur per unit standard and typically includes a nursing visit and a doctor visit within 2-3 days of discharge. Additionally, caregivers will be contacted via telephone within 2 days to answer any questions or address any concerns pertaining to apneic events, home monitor use, or caffeine therapy. Follow up in the pulmonary clinic will be arranged at 42-43 weeks gestational age at which time caregivers will be taught to determine the baseline frequency of monitor alarms on caffeine. At 43 weeks corrected gestational age, caregivers will be instructed to discontinue caffeine therapy and advised to contact the pulmonary clinic should alarm frequency increase. An outpatient recorded oximetry study will be arranged at least 1 week after discontinuation of caffeine therapy. Home pulse oximetry monitoring will be discontinued if no significant events are recorded. Caregivers will be asked to complete 3 brief questionnaires at enrollment, at 1 month after discontinuation of the home monitor, and at 6 months of age. Each questionnaire will ask about topics such as satisfaction with hospital stay, quality of life, and numbers monitor alarms, acute care visits and/or rehospitalizations.

DETAILED DESCRIPTION:
1. Study Design This is a prospective, randomized study. Our primary objective will be to test the hypothesis that early discharge and outpatient monitoring of late preterm to term infants with apnea of prematurity results in decreased length of hospital stay, is safe and cost effective, and results in improved patient satisfaction, as assessed by the PedsQL questionnaire and Impact on Family Scale.
2. Patient Selection and Inclusion/Exclusion Criteria
3. Description of Study Treatments or Exposures/Predictors The investigators will identify all qualified infants who meet eligibility criteria for enrollment, and will obtain informed consent at that time. Infants will not be randomized until their apnea, bradycardia, and/or oxygen desaturation has been the sole remaining discharge criteria for at least 7 days. Prior to randomization, but after the receipt of written informed consent, the investigators will confirm that the primary clinical team has determined that there are no alternate etiologies for the apnea/bradycardia/desaturation events, based on diagnostic testing or clinical judgment.

   Randomization will be stratified according to gestational age at birth to include two broad categories as follows: 1) late preterm infants who are born between 34 0/7 and 36 6/7 weeks gestation (late preterm infants) and 2) term infants who are born at or greater than 37 0/7 weeks gestation. Our aim will be to recruit at least 5 infants in each treatment arm for both late preterm and full term infants.

   Arm A will include continued inpatient monitoring of apnea, bradycardia, and/or desaturation until an event free period of time (5 days per the current standard of care at each participating institution) has been established and deemed appropriate for discharge home per the discretion of the responsible provider. The protocol described in Arm A is currently utilized as a standard of care for many infants locally and nationally and is the first management option utilized at all participating institutions. Arm B will include the initiation of caffeine treatment once randomization has been established. Per current dosing guideline, patients will receive a one-time loading dose of 20 milligrams per kilogram on day 1 with a daily maintenance dose thereafter of 10 milligrams per kilogram. Monitoring of caffeine drug levels will not be included in our protocol as the safety of caffeine treatment in neonates without laboratory monitoring has been well established. After receiving the loading dose of caffeine, infants will receive continued inpatient monitoring of apnea/bradycardia/desaturation until an event free period of time (3 days per the current standard of care at each participating institution) has been established and deemed appropriate for discharge home per the discretion of the responsible provider. Infants discharged home on caffeine therapy will receive instructions regarding use of a home monitor, with alarms set to alarm for heart rate <80 or > 200 beats per minute, or for oxygen saturation level < 90%. The protocol described in Arm B is currently utilized as a standard of care for many infants locally and nationally as a secondary option after observation alone has resulted in a prolonged inpatient stay due to persistent apnea with all other discharge criteria having been met. In a recent retrospective analysis of home monitor use, the investigators found that 1 in 20 infants with apnea of prematurity were discharge home with a monitor.

   Following discharge home, infants in Arm B will be contacted via telephone within 2 days to answer any questions or address any concerns pertaining to apneic events, home pulse oximeter use, or caffeine therapy. Follow up in the pulmonary clinic will be arranged at 42-43 weeks gestational age at which time caregivers will be taught to determine the baseline frequency of monitor alarms on caffeine. At 43 weeks corrected gestational age, caregivers will be instructed to discontinue caffeine therapy and advised to contact the pulmonary clinic should alarm frequency increase. An outpatient recorded oximetry study will be arranged at least 1 week after discontinuation of caffeine therapy. Home pulse oximetry monitoring will be discontinued if no significant events, as previously defined, are recorded.

   Follow up after discharge in both treatment arms will otherwise proceed per unit protocol and typically consists of a home visiting nurse within 2-3 days of hospital discharge and a primary care provider appointment within 2-3 days of hospital discharge.
4. Data Collection Methods, Assessments, Interventions and Schedule (what assessments performed, how often) For infants in both arms, parents will participate in a structured questionnaire at enrollment, and 1 month after hospital discharge for patients in Arm A and 1 month after discontinuation of home monitor use for patients in Arm B. The investigators will also contact families at 6 months of age to determine rehospitalization rates, and frequency of emergency department visits related to respiratory issues.

ELIGIBILITY:
Our study population will include infants who meet the following criteria: (1) Born at greater than or equal to 34 0/7 weeks gestation; (2) Are assigned a diagnosis of apnea, bradycardia, and/or oxygen desaturations by the primary clinical team; (3) Have met all other discharge criteria (i.e. feeding maturity, temperature regulation, etc.) so that apnea/bradycardia/desaturation remains the final discharge issue.

As our intent will be to study infants for whom hospital stay is prolonged as a result of presumed apnea of prematurity, exclusion criteria will include: (1) comorbidities associated with an increased risk of apnea, including neurologic abnormalities such as congenital CNS malformations, seizures, or intracranial bleeds, anatomic abnormalities of the airway, significant congenital heart disease, residual lung disease requiring respiratory support, infectious disease including sepsis, pneumonia, or meningitis, chromosomal abnormalities, and drug withdrawal; (2) prolonged hospitalization for an indication other than apnea, bradycardia and/or oxygen desaturation such as feeding immaturity, temperature instability, or phototherapy; (3) transfer to an outside hospital; (4) provider concern with caregiver ability to safely operate and comply with home monitor use.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Respiratory Events | Within 6 months of age
  respiratory-related acute care visits, emergency department visits, or rehospitalizations
Parent Quality of Life | Within 6 months of age
  Parent-reported quality of life (PedsQL and Impact on Family Scale)